CLINICAL TRIAL: NCT04914234
Title: Premedication With Atenolol Versus Metoprolol for Controlled Hypotensive Anesthesia During Nasal Surgeries. A Randomized Clinical Trial
Brief Title: Premedication With Atenolol Versus Metoprolol for Controlled Hypotensive Anesthesia During Nasal Surgeries
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Damanhour Teaching Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DTH: 21002
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Hypotension Drug-Induced
Keywords: atenolol; controlled hypotension; metoprolol; nasal surgery
MeSH Terms: conditions — Hypotension | interventions — Atenolol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (n=30) (Active Comparator): Atenolol group
  Interventions: Drug: Atenolol Succinate Oral Tablet
- Group M (n=30) (Active Comparator): Metoprolol group
  Interventions: Drug: Metoprolol Succinate Oral Tablet

INTERVENTIONS:
Drug: Atenolol Succinate Oral Tablet — Atenolol 50 mg
  Other Names: Tenormin tablets
  Arms: Group A (n=30)
Drug: Metoprolol Succinate Oral Tablet — Metoprolol 100 mg
  Other Names: Seloken ZOC tablets
  Arms: Group M (n=30)

SUMMARY:
Objectives: To compare the safety and efficacy of oral atenolol versus oral metoprolol as a premedication for controlled hypotensive anesthesia during nasal surgeries.

Background: Mucosal bleeding is the most frequent complication with nasal surgeries, as it interferes with the optimal visualization of the intranasal anatomy, increases operation time, and consequently increases blood loss. There are several pharmacological and non-pharmacological techniques for the appropriate control of intraoperative bleeding.

Patients and Methods: This was a prospective, randomized, double-blind, phase four, comparative clinical trial; carried out on 60 patients, who were candidates for nasal surgeries under general anesthesia at our hospital. Patients were randomly allocated into two equal groups; group A, received oral atenolol, and group M, received oral metoprolol.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status ≤ II
* Age from 21 to 50 years

Exclusion Criteria:

* ASA physical status > II
* Age < 21 years or > 50 years
* Pregnant women
* Breastfeeding
* Bronchial asthma
* Chronic obstructive pulmonary disease
* Diabetes Mellitus
* Hypertension
* Ischemic heart disease
* Rheumatic heart disease
* Heart failure
* Heart block
* Sick sinus syndrome
* Sinus bradycardia
* Chronic hypotension
* Anemia (Hb < 10 g/dl)
* Renal or hepatic dysfunction
* Central nervous system disease
* Allergic fungal sinusitis
* Patients on beta-blockers
* Alcohol or drug abuse
* Anticoagulation therapy,
* Bleeding diathesis
* Agents influencing autonomic nervous system
* Allergy to the study drugs
* Any contraindication of oral intake

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Mean and Standard deviation of Blood loss (ml)(mean±SD) | 5 minutes after the end of surgery
  Amount of blood loss at the end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Shaat, MD, Principal Investigator — Damanhour Teaching Hospital
Locations (1):
- Damanhour Teaching Hospital, Damanhūr, El-Beheira, Egypt